CLINICAL TRIAL: NCT01870492
Title: Improving Patient Access to Stroke Therapy Study
Acronym: IMPACT
Status: Terminated | Type: Observational
Why Stopped: Principle Investigator relocated to a new institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: 19978
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: IV-tPA; Activase; endovascular therapy
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — Tissue Plasminogen Activator; oxotris(2-pyridylmethyl)amineiron(IV)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute ischemic stroke or TIA: Patients presenting with acute ischemic stroke or transient ischemic attack and underwent treatment using Activase and/or endovascular therapy.
  Interventions: Drug: Activase; Device: Endovascular therapy

INTERVENTIONS:
Drug: Activase — Patients treated with Activase
  Other Names: IV-tPA
Device: Endovascular therapy — Patients treated with endovascular therapy, such as IA-tPA, mechanical thrombectomy, etc for acute ischemic stroke or transient ischemic attack.

SUMMARY:
Limited access is a major hurdle in the treatment of AIS; many hospitals, especially rural hospitals, do not have the infrastructure or medical support to effectively treat AIS patients.5 Failure to recognize the signs and symptoms of stroke by the patient and/or emergency medical services (EMS) is another barrier to the timely treatment of AIS. Several studies, including the Paul Coverdell National Acute Stroke Registry (PCNASR), have reported low rates of adherence to stroke care guidelines, suggesting that many AIS patients do not receive proper treatment according to established guidelines. Thus, there remains an increasing need to assess and address the barriers that prevent patient access to proper AIS treatment.

Annually, approximately 20,000 patients are discharged from Wisconsin hospitals with the diagnosis of stroke and an estimated 4,000 patients die from stroke each year in WI. To date, there have been no statewide studies initiated in Wisconsin to assess the regional barriers to the treatment of AIS patients with thrombolytic or endovascular therapy, and many hospitals do not routinely collect and analyze AIS patient data.

The goal of the Improving Patient Access to Stroke Therapy (IMPACT) pilot study is to engage community hospitals statewide to identify the regional barriers to AIS therapy in WI.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical diagnosis of acute ischemic stroke or transient ischemic attack (TIA)
* ICD-9-CM code indicative of stroke or TIA

Exclusion Criteria:

* Clinical diagnosis of intracerebral hemorrhage or subarachnoid hemorrhage
* Stroke or TIA occurred while patient was hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with an acute ischemic stroke (AIS) or transient ischemic attack (TIA) and meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

PRIMARY OUTCOMES:
Identification of regional pre-hospital, hospital, and community barriers to stroke therapy | At end of study (12 months)

SECONDARY OUTCOMES:
Total number of stroke patients treated with acute stroke therapy | At end of study (12 months)
Total number of stroke patients eligible to receive Activase® versus patients eligible but did not receive Activase® | At end of study (12 months)
Use of endovascular therapy in patients who received Activase® versus patients who did not receive Activase® | At end of study (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Osama O Zaidat, MD, MS, Principal Investigator — Medical College Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States